CLINICAL TRIAL: NCT01193660
Title: Double-blind Randomized Controlled Trial to Evaluate the Efficacy and Safety of a Combination Therapy of Allogenic Umbilical Cord Blood and Erythropoietin for Children With Cerebral Palsy
Brief Title: Allogenic Umbilical Cord Blood and Erythropoietin Combination Therapy for Cerebral Palsy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sung Kwang Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RCTUBSC; PBC09-095 (Other: IRB of CHA Bundang Medical Center)
Record Dates: First submitted 2010-08-29; First posted 2010-09-02 (Estimated); Results first posted 2012-03-01 (Estimated); Last update posted 2020-11-24 (Actual); Status verified 2020-11

CONDITIONS: Cerebral Palsy
Keywords: umbilical cord blood; stem cell; cerebral palsy
MeSH Terms: conditions — Cerebral Palsy | interventions — Erythropoietin; Albumins

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Umbilical Cord Blood & Erythropoietin & Rehabilitation (Experimental): Allogenic umbilical cord blood infusion, erythropoietin injection & active rehabilitation
  Interventions: Biological: Umbilical Cord Blood Infusion; Drug: Erythropoietin Injection; Other: Active Rehabilitation
- Erythropoietin & Rehabilitation (Active Comparator): Erythropoietin injection, active rehabilitation
  Interventions: Drug: Erythropoietin Injection; Other: Active Rehabilitation; Other: Placebo Umbilical Cord Blood
- Only Rehabilitation (Placebo Comparator): Active rehabilitation
  Interventions: Other: Active Rehabilitation; Other: Placebo Umbilical Cord Blood; Other: Placebo Erythropoietin

INTERVENTIONS:
Biological: Umbilical Cord Blood Infusion — The subjects will be undertaken allogeneic umbilical cord blood infusion (total nucleated cells > 3x10^7/kg) intravenously under non-myeloablative immunosuppression (maintaining blood level of cyclosporine as 100-200ng/mL for 1 month).
  Other Names: Donated Umbilical Cord Blood Units from Affiliated Cord Blood Bank
  Arms: Umbilical Cord Blood & Erythropoietin & Rehabilitation
Drug: Erythropoietin Injection — Erythropoietin will be given as the schedule of twice a week for 4 weeks with the dosage of 500 IU/kg for 2 times intravenously and 250 IU/kg subcutaneously for 6 times.
  Other Names: Brand name of Erythropoietin: Espogen (made by LG Life Science)
  Arms: Erythropoietin & Rehabilitation; Umbilical Cord Blood & Erythropoietin & Rehabilitation
Other: Active Rehabilitation — All subjects should participate in active rehabilitation. They received two physical and occupational therapy sessions per day. Post discharge, each participant continued to receive rehabilitation therapy at least 3 days per week for additional 5 months.
Other: Placebo Umbilical Cord Blood — Placebo Umbilical Cord Blood will be given except the Experimental arm. Placebo Umbilical Cord Blood was made using peripheral blood. Participants and Investigators maintained as blind.
  Other Names: Placebo Umbilical Cord Blood that resembles cord blood in appearance was designed; : 1.5 to 3 ml of the subject's own blood was collected and mixed with 15 to 20 ml of albumin.
  Arms: Erythropoietin & Rehabilitation; Only Rehabilitation
Other: Placebo Erythropoietin — Placebo Erythropoietin containing Normal Saline
  Arms: Only Rehabilitation

SUMMARY:
This randomized control study is aimed to determine efficacy of umbilical cord blood and erythropoietin combination therapy for children with cerebral palsy.

DETAILED DESCRIPTION:
Cerebral palsy is a disorder of movement and posture that result from a nonprogressive lesion or injury of the immature brain. It is a leading cause of childhood onset disability through one's life. Umbilical cord blood(UCB) is suggested as therapeutic method for cerebral palsy which resulted from animal studies. Stem cells included in UCB is expected to exert therapeutic efficacy for functional recovery.

It is also suggested that erythropoietin is useful to repair neurological injury in brain. The main mechanism of erythropoietin is supposed to be neuroprotection and neurogenesis which would reinforce the effect of stem cell as well.

Although autologous umbilical cord would be safe, the children who have problems at birth seldom have autologous umbilical cord blood. Allogenic umbilical cord blood might be useful for these children if its effect is approved.

ELIGIBILITY:
Inclusion Criteria:

* Known cerebral palsy
* Willing to comply with all study procedure

Exclusion Criteria:

* High risk of pneumonia or renal function deterioration after using of immunosuppressant
* Presence of known genetic disease
* Possibility of drug hypersensitivity which is related to this study remedy
* History of previous cell therapy
* Poor cooperation of guardian,including inactive attitude for rehabilitation
* Intractable seizure disorder
* Autism

Ages: 10 Months to 10 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 105 (Actual)
Dates: Start 2010-05; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Minyoung Kim, MD, PhD, Study Chair — CHA University
Locations (1):
- CHA Bundang Medical Center, Seongnam-si, Gyeonggi-do, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Enrollment Period: May 31, 2010 through April 9, 2011 All participants were recruited at CHA Bundang Medical Center.
Pre-assignment Details: We tried to recruit 106 subjects. Finally 105 patients were enrolled at the beginning of the overall study and none of the participants were washed out before assignment to groups.
Groups:
- Umbilical Cord Blood & Erythropoietin & Rehabilitation: Allogeneic umbilical cord blood infusion (total nucleated cells > 3x10^7/kg intravenously), Erythropoietin injection (twice a week for 4 weeks with the dosage of 500 IU/kg for 2 times intravenously and 250 IU/kg subcutaneously for 6 times), and active rehabilitation
- Erythropoietin & Rehabilitation: Erythropoietin injection (twice a week for 4 weeks with the dosage of 500 IU/kg for 2 times intravenously and 250 IU/kg subcutaneously for 6 times),and active rehabilitation
Period: Overall Study
Arm/Group | Umbilical Cord Blood & Erythropoietin & Rehabilitation | Erythropoietin & Rehabilitation | Only Rehabilitation
Started | 35 | 36 | 34
Completed | 31 | 33 | 32
Not Completed | 4 | 3 | 2
Not completed — Withdrawal by Subject | 2 | 3 | 1
Not completed — Death | 1 | 0 | 0
Not completed — Physician Decision | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Umbilical Cord Blood & Erythropoietin & Rehabilitation | Erythropoietin & Rehabilitation | Only Rehabilitation | Total
Number analyzed (Participants) | 35 | 36 | 34 | 105
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 35 | 36 | 34 | 105
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 45.71 (18.91) | 50.05 (24.45) | 46.0 (19.58) | 47.30 (21.07)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 11 | 9 | 33
  Male | 22 | 25 | 25 | 72
Region of Enrollment [Number; unit: participants]
  Korea, Republic of | 35 | 36 | 34 | 105

OUTCOME MEASURES:

1. Primary Outcome: Changes in Motor Performance
Description: GMPM (Gross Motor Performance Measure) as a standardized measurement tool for assessing quality of movement regarding 3 properties of 5 ones; alignment, coordination, dissociated movement, stability, and weight shift (range: 0~100, Higher value means better motor quality). We reported changes of GMPM score between each assessment time points. Categories of outcome table are baseline and values of just subtracting the latter raw scores from the former ones.
Time Frame: Baseline -1 month - 3 months - 6 months
Population: Intention to treat
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Umbilical Cord Blood & Erythropoietin & Rehabilitation | Erythropoietin & Rehabilitation | Only Rehabilitation
Number analyzed (Participants) | 31 | 33 | 32
units on a scale
  Baseline | 34.5 (2.7) | 38.2 (2.8) | 35.5 (2.9)
  1 month - Baseline | 7.00 (1.3) | 4.5 (0.6) | 6.0 (1.0)
  3 months - Baseline | 11.5 (1.5) | 7.5 (0.8) | 8.1 (1.2)
  6 months - Baseline | 14.5 (1.8) | 9.2 (0.8) | 9.6 (1.2)
  3 months - 1 month | 4.5 (0.7) | 2.9 (0.5) | 2.1 (0.6)
  6 months - 1 month | 7.5 (0.9) | 4.7 (0.7) | 3.6 (0.7)
  6 months - 3 months | 3.1 (0.6) | 1.7 (0.5) | 1.5 (0.4)
Statistical Analysis 1: Comparison: Umbilical Cord Blood & Erythropoietin & Rehabilitation vs Erythropoietin & Rehabilitation vs Only Rehabilitation; In our analysis, the null hypothesis is that the effects of 3 experimental groups are same, and the alternative hypothesis is that the therapeutic effect of combination intervention Group (Umbilical Cord Blood + Erythropoietin + Rehabilitation) is higher than that of either Erythropoietin + Rehabilitation or Rehabilitation Group. This is a pilot study and power calculation was not applicable. The sample size of each group is over 30 and is considered to follow approximately normal distribution; Test type: Superiority or Other; p < 0.05, Repeated Measure ANOVA; Wilks' Lambda (group*visit effect) = 2.59

2. Secondary Outcome: Changes in Cognitive Neurodevelopmental Outcome
Description: Korean version of Bayley Scale of Infant Development-II (K-BSID-II) Mental Scales (higher value means better mental function: 0 - worst, 178 - best). We reported changes of BSID-II Mental Scale raw score between each assessment time points. Categories of outcome data are values of subtracting the latter scores from the former ones.
Time Frame: Baseline -1 month - 3 months - 6 months
Population: Intention to treat
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Umbilical Cord Blood & Erythropoietin & Rehabilitation | Erythropoietin & Rehabilitation | Only Rehabilitation
Number analyzed (Participants) | 31 | 33 | 32
units on a scale
  BSID-II Mental Scale: Baseline | 94.1 (9.1) | 105.9 (8.9) | 86.6 (9.0)
  BSID-II Mental Scale: 1 month - Baseline | 8.2 (1.3) | 3.4 (0.5) | 3.3 (0.6)
  BSID-II Mental Scale: 3 months - Baseline | 12.0 (1.4) | 7.4 (0.9) | 5.8 (0.8)
  BSID-II Mental Scale: 6 months - Baseline | 17.6 (1.8) | 11.5 (1.3) | 9.9 (1.6)
  BSID-II Mental Scale: 3 months - 1 month | 3.8 (0.8) | 4.0 (0.7) | 2.5 (0.7)
  BSID-II Mental Scale: 6 months - 1 month | 9.4 (1.4) | 8.1 (1.3) | 6.6 (1.4)
  BSID-II Mental Scale: 6 months - 3 months | 5.6 (1.2) | 4.1 (0.8) | 4.1 (1.0)
Statistical Analysis 1: Comparison: Umbilical Cord Blood & Erythropoietin & Rehabilitation vs Erythropoietin & Rehabilitation vs Only Rehabilitation; The null hypothesis is that in terms of K-BSID-II MENTAL Scale, the effects of 3 groups are same, and the alternative one is that the therapeutic effect of combination intervention Group (Umbilical Cord Blood + Erythropoietin + Rehabilitation) is higher than that of either Erythropoietin + Rehabilitation or Rehabilitation Group. This is a pilot study and power calculation was not applicable. The sample size of each group is over 30 and is considered to follow approximately normal distribution; Test type: Superiority or Other; p < 0.05, Repeated Measure ANOVA; Wilks' Lambda (group*visit effect) = 3.94

3. Secondary Outcome: Changes in Motor Neurodevelopmental Outcome
Description: Korean version of Bayley Scale of Infant Development-II (K-BSID-II) Motor Scales (higher value means better motor function: 0 - worst, 111 - best). We reported changes of BSID-II Motor Scale raw score between each assessment time points. Categories of outcome data are values of subtracting the latter scores from the former ones.
Time Frame: Baseline - 1 month - 3 months - 6 months
Population: Intention to treat
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Umbilical Cord Blood & Erythropoietin & Rehabilitation | Erythropoietin & Rehabilitation | Only Rehabilitation
Number analyzed (Participants) | 31 | 33 | 32
units on a scale
  BSID-II Motor Scale: Baseline | 45.2 (4.7) | 53.3 (5.0) | 45.5 (4.6)
  BSID-II Motor Scale: 1 month - Baseline | 5.0 (1.5) | 5.2 (2.1) | 2.7 (0.6)
  BSID-II Motor Scale: 3 months - Baseline | 9.5 (1.9) | 6.8 (2.1) | 4.3 (0.8)
  BSID-II Motor Scale: 6 months - Baseline | 11.7 (2.0) | 7.6 (2.2) | 5.2 (0.9)
  BSID-II Motor Scale: 3 months - 1 month | 4.5 (1.0) | 1.6 (0.5) | 1.5 (0.4)
  BSID-II Motor Scale: 6 months - 1 month | 6.7 (1.3) | 2.5 (0.6) | 2.5 (0.5)
  BSID-II Motor Scale: 6 months - 3 months | 2.2 (0.6) | 0.9 (0.4) | 1.0 (0.4)
Statistical Analysis 1: Comparison: Umbilical Cord Blood & Erythropoietin & Rehabilitation vs Erythropoietin & Rehabilitation vs Only Rehabilitation; The null hypothesis is that in terms of K-BSID-II MOTOR Scale, the effects of 3 groups are same, and the alternative one is that the therapeutic effect of combination intervention Group (Umbilical Cord Blood + Erythropoietin + Rehabilitation) is higher than that of either Erythropoietin + Rehabilitation or Rehabilitation Group. This is a pilot study and power calculation was not applicable. The sample size of each group is over 30 and is considered to follow approximately normal distribution; Test type: Superiority or Other; p < 0.05, Repeated Measure ANOVA; Wilks' Lambda (group*visit effect) = 2.70

4. Secondary Outcome: Changes in Brain MRI
Description: Changes on brain Diffusion Tensor Image (DTI); DTI provides quantitative information about the microscopic integrity of white matter. White matter normally possesses a high degree of diffusion anisotropy than gray matter. We can measure fractional anisotropy (FA) value in DTI imaging and it ranges from 0 to 1. Higher FA value of a certain region of interest means the area has more integrity of white matter.
Time Frame: Baseline - 6 months
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Umbilical Cord Blood & Erythropoietin & Rehabilitation | Erythropoietin & Rehabilitation | Only Rehabilitation
Number analyzed (Participants) | 30 | 31 | 29
units on a scale
  Anterior portion of Rt. posterior Internal Capsule | 0.03 (0.01) | 0.01 (0.01) | 0.01 (0.01)
  Posterior portion of Rt posterior Internal Capsule | 0.04 (0.01) | 0.02 (0.01) | 0.02 (0.02)
  Anterior portion of Lt. posterior Internal Capsule | 0.03 (0.01) | 0.02 (0.01) | 0.04 (0.02)
  Posterior portion of Lt posterior Internal Capsule | 0.05 (0.02) | 0.04 (0.02) | 0.05 (0.02)

5. Secondary Outcome: Comparison of Changes in Brain Glucose Metabolism Using by Brain 18F-FDG PET: Increased and Decreased Areas of Brain Glucose Metabolism
Description: 18F-FDG PET imaging was performed twice prior to and then 2 weeks post-treatment. Ninety slices of each emission image were obtained, and all scans were reviewed by a nuclear physician. Spatial pre-processing and statistical analyses were performed using SPM8 implanted in Matlab to compare differences in regional brain glucose metabolism between groups and differences between pre- and post-therapy imaging data. We reported increased areas and decreased areas of glucose metabolism in three groups. We defined that "1" refers to INCREASED areas, "-1", DECREASED areas and "0", just NO CHANGE.
Time Frame: Baseline - 2 weeks
Population: Intention to treat
Measure: Number; unit: units on a scale
Arm/Group | Umbilical Cord Blood & Erythropoietin & Rehabilitation | Erythropoietin & Rehabilitation | Only Rehabilitation
Number analyzed (Participants) | 31 | 33 | 32
units on a scale
  Rt. Lentiform Nucleus, Gray Matter, Putamen | 1 | 0 | 0
  Lt. Frontal Lobe, Medial Frontal Gyrus | 1 | 0 | 0
  Lt. Sub-lobar, Insula | 1 | 0 | -1
  Lt. Lentiform Nucleus, Gray Matter, Putamen | 1 | 0 | 0
  Lt.Lentiform Nucleus, Gray Matter, Globus Pallidus | 1 | 0 | 0
  Lt. Midbrain (Thalamus) | 1 | 0 | 0
  Rt. Parietal Lobe, Precuneus | 1 | 0 | 0
  Lt. Temporal Lobe, Middle Temporal Gyrus | 1 | 0 | -1
  Rt. Parietal Lobe, Pre- and Post-central Gyrus | 1 | 0 | 0
  Rt. Frontal Lobe, Paracentral Lobule | 0 | 1 | 0
  Rt. Limbic Lobe, Anterior Cingulate | 0 | 1 | 0
  Lt. Frontal Lobe, Precentral Gyrus | 0 | 1 | 0
  Lt. Lentiform Nucleus, Putamen | 0 | 1 | 0
  Rt. Cerebellar Anterior Lobe, Culmen | 0 | 1 | 1
  Lt. Cerebellar Posterior Lobe, Cerebellar Tonsil | 0 | 1 | 1
  Rt. Frontal Lobe, Orbital Gyrus | 0 | 1 | 1
  Rt. Occipital Lobe, Middle Occipital Gyrus | -1 | 0 | 0
  Lt. Limbic Lobe, Parahippocampal Gyrus | -1 | 0 | 0
  Rt. Limbic Lobe, Parahippocampal Gyrus | -1 | 0 | -1
  Rt Cerebellum, Posterior Lobe, Declive | 0 | -1 | 0
  Rt Cerebellum, Anterior Lobe, Culmen, Occipital | 0 | -1 | 0
  Lt Cerebellum, Posterior Lobe, Declive, Occipital | 0 | -1 | 0
  Lt. Frontal Lobe, Middle Frontal Gyrus | 0 | 0 | -1
  Rt. Frontal Lobe, Middle Frontal Gyrus | 0 | 0 | -1
  Rt. Frontal Lobe, Sub-gyral | 0 | 0 | -1
  Lt. Temporal Lobe, Fusiform Gyrus | 0 | 0 | -1
  Lt. Temporal Lobe, Inferior Temporal Gyrus | 0 | 0 | -1
  Rt. Temporal Lobe, Middle Temporal Gyrus | 0 | 0 | -1
Statistical Analysis 1: Comparison: Umbilical Cord Blood & Erythropoietin & Rehabilitation vs Erythropoietin & Rehabilitation vs Only Rehabilitation; In our analysis, the null hypothesis is that the effects of three experimental groups are same each other, and the alternative hypothesis is that the therapeutic effect of combination intervention Group (Umbilical Cord Blood + Erythropoietin + Rehabilitation) has much higher than that of either Erythropoietin + Rehabilitation Group or Rehabilitation Group. This study is a pilot study and therefore, power calculation was not applicable in our study. The sample size of each group is more than 30; Test type: Superiority or Other; p = 0.05, t-test, 2 sided — The baseline and post-therapy data of each group were compared using paired t-test statistics; Voxels with an uncorrected p-value of <0.05 were considered significant, and an extent threshold Ke of 100 voxels was set by SPM implanted in Matlab

6. Secondary Outcome: Changes in Functional Performance in Daily Activities
Description: Pediatric Evaluation of Disability Inventory (PEDI) for assessing functional performance in daily activities in children (All values are adjusted and higher value means better functional performance, 0 - worst, 100 - best). We reported here 2 scales and 3 domains of each scale: a Functional Skill Scale (FSS) and a Caregiver Assistance Scale (CAS) which are divided respectively into 3 domains: self care, mobility, and social function. Categories of outcome table are each domain scores measured at each assessment time point.
Time Frame: Baseline -1 month - 3 months - 6 months
Population: Intention to treat
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Umbilical Cord Blood & Erythropoietin & Rehabilitation | Erythropoietin & Rehabilitation | Only Rehabilitation
Number analyzed (Participants) | 31 | 33 | 32
units on a scale
  Self care of FSS: Baseline | 39.1 (2.5) | 38.2 (2.7) | 37.4 (2.2)
  Self care of FSS: 1 month | 42.2 (2.2) | 40.4 (2.9) | 40.0 (2.2)
  Self care of FSS: 3 months | 44.7 (2.4) | 43.5 (2.9) | 41.7 (2.3)
  Self care of FSS: 6 months | 46.5 (2.5) | 45.0 (2.8) | 42.8 (2.3)
  Mobility of FSS: Baseline | 24.8 (3.7) | 29.2 (4.3) | 24.9 (3.7)
  Mobility of FSS: 1 month | 28.1 (3.9) | 32.4 (4.3) | 27.9 (3.8)
  Mobility of FSS: 3 months | 31.7 (4.3) | 34.6 (4.3) | 29.3 (3.9)
  Mobility of FSS: 6 months | 34.6 (4.3) | 36.6 (4.4) | 31.4 (3.9)
  Social function of FSS: Baseline | 40.0 (3.5) | 40.1 (3.3) | 34.8 (3.5)
  Social function of FSS: 1 month | 42.8 (3.6) | 42.5 (3.3) | 37.5 (3.6)
  Social function of FSS: 3 months | 46.4 (3.9) | 45.8 (3.3) | 40.0 (3.5)
  Social function of FSS: 6 months | 49.1 (3.6) | 47.8 (3.4) | 42.3 (3.9)
  Self care of CAS: Baseline | 18.0 (4.1) | 17.9 (3.7) | 15.3 (3.2)
  Self care of CAS: 1 month | 20.1 (4.0) | 21.1 (3.8) | 19.0 (3.7)
  Self care of CAS: 3 months | 27.0 (4.3) | 24.2 (3.9) | 21.5 (3.7)
  Self care of CAS: 6 months | 29.4 (4.0) | 26.0 (4.1) | 23.1 (3.9)
  Mobility of CAS: Baseline | 14.6 (4.1) | 19.7 (4.8) | 13.5 (4.0)
  Mobility of CAS: 1 month | 19.6 (4.5) | 22.6 (4.9) | 15.6 (4.2)
  Moblity of CAS: 3 months | 22.5 (5.1) | 26.0 (5.3) | 19.3 (4.5)
  Mobility of CAS: 6 months | 24.9 (5.5) | 29.2 (5.4) | 24.0 (4.8)
  Social function of CAS: Baseline | 23.0 (5.2) | 24.7 (3.9) | 18.2 (4.4)
  Social function of CAS: 1 month | 28.5 (5.6) | 30.0 (4.5) | 21.1 (4.8)
  Social function of CAS: 3 months | 34.8 (6.0) | 34.2 (4.8) | 24.2 (5.0)
  Social function of CAS: 6 months | 38.4 (6.2) | 36.2 (4.6) | 27.6 (5.3)

7. Primary Outcome: Changes in Standardized Gross Motor Function
Description: GMFM (Gross Motor Function Measure) as a standardized measurement tool for assessing Gross Motor Function consisting of sub-scales; lying & rolling, sitting, crawling & kneeling, standing, walking, running & jumping (range: 0~100 , Higher value means better gross motor function). We reported changes of GMFM between each assessment time points. Categories of outcome table are baseline and values of just subtracting the latter raw scores from the former ones.
Time Frame: Baseline - 1 month - 3 months - 6 months
Population: Intention to treat
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Umbilical Cord Blood & Erythropoietin & Rehabilitation | Erythropoietin & Rehabilitation | Only Rehabilitation
Number analyzed (Participants) | 31 | 33 | 32
units on a scale
  Baseline | 36.0 (4.7) | 42.6 (4.9) | 36.8 (4.5)
  1 month - Baseline | 3.7 (0.4) | 4.3 (0.5) | 4.6 (0.6)
  3 months - Baseline | 6.5 (0.9) | 6.8 (0.8) | 6.4 (0.7)
  6 months - Baseline | 9.1 (1.2) | 9.0 (1.1) | 7.8 (0.9)
  3 months - 1 month | 2.9 (0.8) | 2.5 (0.5) | 1.8 (0.4)
  6 months - 1 month | 5.4 (1.2) | 4.7 (0.9) | 3.1 (0.6)
  6 months - 3 months | 2.6 (0.5) | 2.2 (0.6) | 1.3 (0.4)
Statistical Analysis 1: Comparison: Umbilical Cord Blood & Erythropoietin & Rehabilitation vs Erythropoietin & Rehabilitation vs Only Rehabilitation; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, Repeated Measure ANOVA; interaction of group and visit = 0.90

8. Secondary Outcome: Changes in Functional Independence in Daily Activities
Description: WeeFIM (Functional Independence Measure for Children) measures functional independence in daily activities. WeeFIM contains 18 items and each item is ranked from complete dependence (scored as 1) to complete independence (scored as 7). The range is from 18 to 126 and higher scores mean more independent performance in daily activities. Categories of outcome table are total WeeFIM scores measured at each assessment time point.
Time Frame: Baseline - 1 month - 3 months - 6 months
Population: Intention to treat
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Umbilical Cord Blood & Erythropoietin & Rehabilitation | Erythropoietin & Rehabilitation | Only Rehabilitation
Number analyzed (Participants) | 31 | 33 | 32
units on a scale
  Baseline | 34.1 (3.8) | 36.6 (3.7) | 31.4 (2.9)
  1 month | 35.6 (4.1) | 37.5 (3.8) | 33.2 (3.1)
  3 months | 38.7 (4.7) | 38.5 (4.1) | 37.1 (3.8)
  6 months | 41.1 (4.8) | 40.3 (4.2) | 37.7 (4.1)
Statistical Analysis 1: Comparison: Umbilical Cord Blood & Erythropoietin & Rehabilitation vs Erythropoietin & Rehabilitation vs Only Rehabilitation; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, Repeated Measure ANOVA; Wilks' Lambda (group*visit effect) = 1.279

9. Secondary Outcome: Changes in Muscle Strength
Description: Summation of MMT (manual muscle strength test score): summated scores of the manual muscle strength test (zero=0, trace=1, poor=2, fair=3, good=4, normal=5) for flexors, extensors, abductors, and adductors of bilateral shoulder and hip joints; flexors and extensors of bilateral elbow, wrist, and knee; dorsiflexors and plantar flexors of the ankles (range: 0 ~ 160) Higher score means better muscle strength. Categories of outcome table are summation of MMT scores measured at each assessment time point.
Time Frame: Baseline - 1 month - 3 months - 6 months
Population: Intention to treat
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Umbilical Cord Blood & Erythropoietin & Rehabilitation | Erythropoietin & Rehabilitation | Only Rehabilitation
Number analyzed (Participants) | 31 | 33 | 32
units on a scale
  Baseline | 100.7 (5.5) | 104.8 (4.4) | 100.3 (4.6)
  1 month | 105.0 (4.9) | 106.8 (4.5) | 101.8 (4.6)
  3 months | 107.8 (4.4) | 107.7 (4.5) | 103.6 (4.6)
  6 months | 109.9 (4.6) | 109.3 (4.5) | 104.3 (4.6)
Statistical Analysis 1: Comparison: Umbilical Cord Blood & Erythropoietin & Rehabilitation vs Erythropoietin & Rehabilitation vs Only Rehabilitation; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, Repeated Measure ANOVA; Wilks' Lambda (group*visit effect) = 0.996

10. Secondary Outcome: Changes in Hand Function
Description: QUEST (Quality of Upper Extremity Skills Test) as a standardized measurement tool for assessing hand function consisting of sub-scales; dissociated movement, grasps, weight bearing, and protective extension. These are standardized to range from zero (or below zero in grasp section) to 100 and higher values mean better hand function. We reported QUEST differences between each assessment times.
Time Frame: Baseline - 1 month - 3 months - 6 months
Population: Intention to treat
Measure: Mean (Standard Error); unit: units on a scale
Arm/Group | Umbilical Cord Blood & Erythropoietin & Rehabilitation | Erythropoietin & Rehabilitation | Only Rehabilitation
Number analyzed (Participants) | 31 | 33 | 32
units on a scale
  Baseline | 36.0 (6.4) | 52.8 (4.9) | 43.0 (5.5)
  1 month - Baseline | 5.0 (1.4) | 5.7 (1.7) | 6.6 (1.4)
  3 months - Baseline | 11.1 (2.2) | 8.8 (2.0) | 10.5 (1.8)
  6 months - Baseline | 13.9 (2.6) | 10.7 (2.2) | 13.0 (2.4)
  3 months - 1 month | 5.7 (1.6) | 3.1 (1.0) | 3.5 (1.7)
  6 months - 1 month | 8.4 (2.0) | 5.1 (1.3) | 6.4 (2.1)
  6 months - 3 months | 2.8 (0.8) | 2.4 (0.8) | 3.1 (1.2)
Statistical Analysis 1: Comparison: Umbilical Cord Blood & Erythropoietin & Rehabilitation vs Erythropoietin & Rehabilitation vs Only Rehabilitation; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, Repeated Measure ANOVA; Wilks' Lambda (group*visit effect) = 0.56

11. Secondary Outcome: Number of Participants With Serious Adverse Events as a Measure of Safety,Which Are Related to Umbilical Cord Blood, Erythropoietin, or Immunosuppressant
Description: The number of patients with serious adverse events within each group; Serious adverse events were defined as any event that resulted in death, was life-threatening, required hospitalization or prolonged the hospital stay, or was otherwise serious in the judgment of the investigator.
Time Frame: 6 months
Measure: Number; unit: participants
Arm/Group | Umbilical Cord Blood & Erythropoietin & Rehabilitation | Erythropoietin & Rehabilitation | Only Rehabilitation
Number analyzed (Participants) | 31 | 33 | 32
participants | 3 | 3 | 3
Statistical Analysis 1: Comparison: Umbilical Cord Blood & Erythropoietin & Rehabilitation vs Erythropoietin & Rehabilitation vs Only Rehabilitation; Test type: Superiority or Other; p < 0.05, Fisher Exact; We compared the ratio of participants with a certain adverse event (AE) and without the AE between three groups using Fisher Exact test

ADVERSE EVENTS:
Time Frame: Baseline - 1 month - 3 months - 6 months
Arm/Group | Umbilical Cord Blood & Erythropoietin & Rehabilitation | Erythropoietin & Rehabilitation | Only Rehabilitation
Serious Adverse Events (participants affected / at risk) | 3/35 | 3/6 | 3/8
Other Adverse Events (participants affected / at risk) | 30/35 | 29/36 | 32/34
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Umbilical Cord Blood & Erythropoietin & Rehabilitation (N=35) | Erythropoietin & Rehabilitation (N=6) | Only Rehabilitation (N=8)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (3) | 1 (1)
Seizure (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Influenza (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 1 (1)
Death (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) — One death at 14 wks post-transplantation. She was a 25 mo-old with spastic quadriplegia from profound hypoxia. She was unable to control her head and showed poor oral function. She had been medically stable. The cause was supposed to be suffocation.
Urinary tract infection (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Umbilical Cord Blood & Erythropoietin & Rehabilitation (N=35) | Erythropoietin & Rehabilitation (N=36) | Only Rehabilitation (N=34)
Seizure (Nervous system disorders) | 1 (1) | 3 (6) | 3/18 (7)
Febrile convulsioin (Nervous system disorders) | 2 (3) | 1/14 (1) | 0/18 (0)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 4/14 (4) | 3/18 (3)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 0/14 (0) | 0/18 (0)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 18 (20) | 19 (23) | 21 (24)
Herpangina (Infections and infestations) | 0 (0) | 2/14 (2) | 1/18 (1)
Constipation (Gastrointestinal disorders) | 5 (5) | 4/14 (4) | 5/18 (5)
Dyspepsia (Gastrointestinal disorders) | 5 (5) | 2 (2) | 2/18 (2)
Nausea, vomiting (Gastrointestinal disorders) | 6 (6) | 5 (5) | 2/18 (2)
Diarrhea (Gastrointestinal disorders) | 6 (6) | 2 (2) | 2/18 (2)
Colitis (Gastrointestinal disorders) | 0 (0) | 1/14 (1) | 2/18 (2)
Anorexia (Gastrointestinal disorders) | 5 (5) | 2 (2) | 1/18 (1)
Dermatitis (Skin and subcutaneous tissue disorders) | 0 (0) | 2 (2) | 2/18 (2)
Urticaria (Skin and subcutaneous tissue disorders) | 2 (2) | 1/14 (1) | 4/18 (4)
Hirsuitism (Skin and subcutaneous tissue disorders) | 2 (2) | 0/0 (0) | 0/0 (0)
Alopecia (Skin and subcutaneous tissue disorders) | 1 (1) | 0/0 (0) | 0/0 (0)
Irritability (Psychiatric disorders) | 4 (4) | 0/14 (0) | 0/18 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 1 (1) | 1/18 (1)
Otitis media acute (Ear and labyrinth disorders) | 1 (1) | 1/14 (1) | 0/18 (0)
Conjunctival irritations (Eye disorders) | 0 (0) | 1/14 (1) | 1/18 (2)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 0/0 (0) | 0/18 (0)
Fever (Infections and infestations) | 12 (12) | 4 (4) | 8/18 (8)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 3 (3) | 1 (1) | 1/18 (1) — Temporary O2 desaturation(89-91%) at the end of UCB infusion in UCB group; O2 desaturation(91%) shortly during sedation for PET in EPO group; O2 desaturation(71-95%) intermittently during 47 min maybe from postictal respiratory depression in control

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes